CLINICAL TRIAL: NCT01472029
Title: Multicenter, Explorative Phase II Study of Perioperative 5-FU, Leucovorin, Docetaxel, and Oxaliplatin (FLOT) in Combination With Trastuzumab in Patients With HER2-positive, Locally Advanced, Resectable Adenocarcinoma of the Gastroesophageal Junction or Stomach (HerFLOT)
Brief Title: Explorative Phase II Study of Perioperative Treatment in Patients With Adenocarcinoma of the Gastroesophageal Junction or Stomach
Acronym: HerFLOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-STO-0310; 2011-001507-13 (EudraCT Number)
Record Dates: First submitted 2011-10-24; First posted 2011-11-16 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Adenocarcinoma of the Stomach
Keywords: Adenocarcinoma; Gastroesophageal junction; Stomach; HER2
MeSH Terms: conditions — Adenocarcinoma | interventions — Fluorouracil; Leucovorin; Docetaxel; Oxaliplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT), trastuzumab (Experimental)
  Interventions: Drug: 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT), trastuzumab; Drug: Post-operative treatment trastuzumab mono therapy

INTERVENTIONS:
Drug: 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT), trastuzumab — Pre-operative treatment 4 cycles and post-operative treatment 4 cycles:
  Trastuzumab 4 mg/kg BW (6 mg loading dose at 1st administration), iv over 1 h on day 1 of each 14 day cycle
  Docetaxel 50 mg/m², iv over 2 h on day 1 of each 14 day cycle
  Oxaliplatin 85 mg/m² in 500 ml G5%, iv over 2h on day 1 of each 14 day cycle
  Leucovorin 200 mg/m² in 250 ml NaCl 0,9%, iv over 1 h on day 1 of each cycle
  5-FU 2600 mg/m², iv over 24 h on day 1 of each 14 day cycle
Drug: Post-operative treatment trastuzumab mono therapy — Trastuzumab mono therapy for 9 cycles:
  Trastuzumab 6 mg/kg BW, iv over 1 h on day 1 of each 21 day cycle

SUMMARY:
The purpose of this study is to determine the rate of complete pathological responses (percentage of patients with pCR referring to the total number of enrolled and eligible patients), as evaluated centrally by a reference pathologist.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed adenocarcinoma of the gastroesophageal junction (AEG I-III) or the stomach (uT2, uT3, uT4, any N category, M0), or any T N+ M0 patient, with the following specifications: Endosonography and an esophageal-gastro-duodenoscopy; Categorization of gastroesophageal junction tumors according to the classification by Siewert (1987, cf. appendix 2)

* Detection of an adenocarcinoma with HER2 3+ (IHC) or HER2 2+ (IHC) with amplification proven by FISH, SISH or CISH by an accredited local pathologist (for quality assurance tumor samples have to be available for a subsequent central review)
* No preceding cytotoxic or targeted therapy
* Male and female patients aged ≥ 18 years. If able to reproduce, patients must be willing to use highly effective methods of contraception during treatment and for 6 months after the end of treatment (adequate: methods fulfilling the requirements of the Note for guidance on non-clinical safety studies for the conduct of human clinical trials for pharmaceuticals [CPMP/ICH/286/95 mod]). Female patients with reproductive ability must have performed a negative pregnancy test within 7 days of study entry.
* ECOG ≤ 2
* Exclusion of distant metastasis by CT of thorax and abdomen, bone scan or MRI (if osseous lesions are suspected due to clinical signs)
* Laparoscopic exclusion of peritoneal carcinomatosis, if suspected clinically
* Adequate haematological, hepatic and renal function parameters: Leukocytes ≥ 3000/mm³, platelets ≥ 100,000/mm3; Serum creatinine ≤ 1.5 x upper limit of normal, or GFR > 40 ml/min; Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.5 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal
* Normal cardiac ejection fraction, as assessed by echocardiography
* Written patient consent form

Exclusion Criteria:

* Known hypersensitivity against trastuzumab, murine proteins, 5-FU, leucovorin, oxaliplatin or docetaxel
* Other known contraindications against trastuzumab, 5-FU, leucovorin, oxaliplatin, or docetaxel
* Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV
* Clinically significant valvular defect
* Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
* Known brain metastases
* Severe dyspnoea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy
* Other severe internal disease or acute infection
* Peripheral polyneuropathy > NCI Grade II
* Chronic inflammatory bowel disease
* On-treatment participation in another clinical study in the period 30 days prior to inclusion and during the study
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
* Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
* Any other concurrent antineoplastic treatment including irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08-25 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
Rate of complete pathological responses (percentage of patients with pCR referring to the total number of enrolled and eligible patients), as evaluated centrally by a reference pathologist. | From enrollment to surgery after pre-operative treatment (4 cycles = 8 weeks) for 9 weeks.
  The experimental therapy would be rated as insufficiently active, if the observed pCR rate is 10 % or lower, as this corresponds to the expectations after chemotherapy alone.
  The experimental therapy would be considered to be a promising candidate for further development (e.g. in a phase III trial), if the true pCR rate amounted to 20% or more.

SECONDARY OUTCOMES:
R0 resection rate | From enrollment to surgery after pre-operative treatment (4 cycles = 8 weeks) for 9 weeks.
  The R0 rate is defined as the number of patients with negative surgical margins and no tumor left macroscopically, divided by the total number of recruited eligible patients.
Relapse-free survival | From enrollment to end of follow up assessed up to 58 months
  Relapse-free survival (RFS) will be defined as the time from enrolment to the time of disease progression or relapse or death, or to the date of last tumor assessment without any such event (censored observation)
Overall survival | From enrollment to end of follow up assessed up to 58 months.
  The duration of overall survival (OS) will be determined by measuring the time interval from enrolment to the date of death or last observation, including survival rates after 1, 2 and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf D Hofheinz, Prof. Dr., Principal Investigator — Tagestherapiezentrum am ITM & III. Medizinische Klinik, Universitätsmedizin Mannheim, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim
Locations (1):
- Tagestherapiezentrum am ITM & III. Medizinische Klinik Universitätsmedizin Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Hofheinz RD, Hegewisch-Becker S, Kunzmann V, Thuss-Patience P, Fuchs M, Homann N, Graeven U, Schulte N, Merx K, Pohl M, Held S, Keller R, Tannapfel A, Al-Batran SE. Trastuzumab in combination with 5-fluorouracil, leucovorin, oxaliplatin and docetaxel as perioperative treatment for patients with human epidermal growth factor receptor 2-positive locally advanced esophagogastric adenocarcinoma: A phase II trial of the Arbeitsgemeinschaft Internistische Onkologie Gastric Cancer Study Group. Int J Cancer. 2021 Sep 15;149(6):1322-1331. doi: 10.1002/ijc.33696. Epub 2021 May 29. PMID 34019698